CLINICAL TRIAL: NCT06286020
Title: A Randomized Controlled Study to Explore the Effect of Virtual Reality Therapy on Dysphagia in Wallenberg Syndrome
Brief Title: Effect of Virtual Reality Therapy on Dysphagia in Wallenberg Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR-Zhenqiu
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Wallenberg Syndrome
MeSH Terms: conditions — Lateral Medullary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): conventional dysphagia treatment and Virtual Reality Therapy are provided
  Interventions: Device: Virtual Reality Therapy; Behavioral: Conventional dysphagia treatment
- The control group (Active Comparator): conventional dysphagia treatment is provided
  Interventions: Behavioral: Conventional dysphagia treatment

INTERVENTIONS:
Device: Virtual Reality Therapy — The therapist begins by assessing the patient's swallowing abilities and creating a personalized treatment plan. This involves determining the appropriate Virtual Reality Therapy scenarios, difficulty levels, and specific swallowing goals tailored to the patient's condition.
  Arms: The experimental group
Behavioral: Conventional dysphagia treatment — Conventional dysphagia treatment included oropharyngeal muscle movement training, orofacial alternating hot and cold stimulation, Masako swallowing training, Mendelsohn maneuver, therapeutic ingestion training, intermittent oral-esophageal tube feeding, etc., 30 min each time, once a day for 14 consecutive days.

SUMMARY:
The goal of this clinical trial is to learn about on dysphagia in wallenberg syndrome. The main questions it aims to answer are:

the efficacy of Virtual Reality Therapy in the rehabilitation of patients with dysphagia in Wallenberg syndrome.

Participants received conventional dysphagia treatment and Virtual Reality Therapy once a day for 14 days. Researchers compared the control group to see the effect and mechanism of Virtual Reality Therapy.

DETAILED DESCRIPTION:
Virtual Reality technology has revolutionized various fields, and its application in rehabilitation medicine is particularly noteworthy. Virtual Reality provides immersive environments that simulate real-life situations, making it an invaluable tool in the rehabilitation process.

The goal of this clinical trial is to learn about on dysphagia in wallenberg syndrome. The main questions it aims to answer are:

the efficacy of Virtual Reality Therapy in the rehabilitation of patients with dysphagia in Wallenberg syndrome.

Participants received conventional dysphagia treatment and Virtual Reality Therapy once a day for 14 days. Researchers compared the control group to see the effect and mechanism of Virtual Reality Therapy.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 18-85 years and right-handed;
* first onset, vital signs stable and conscious;
* the dysphagia confirmed by videofluoroscopic swallowing study;
* no cognitive impairment, the mini-mental state examination score: >17 for those with an illiterate education, >20 for those with an elementary education, and >24 for those with a secondary education and above;
* cranial integrity without craniotomy and/or craniectomy;
* patient and/or his/her relative agrees and signs written informed consent.

Exclusion Criteria:

* combined ischemic foci at other sites;
* presence of organic swallowing dysfunction or pre-existing dysphagia due to Parkinson's disease, dementia, and others;
* severe cardiac, pulmonary, hepatic, and renal insufficiency and vital organ failure;
* infected or broken skin on the head;
* poorly controlled epilepsy;
* poor patient compliance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
standardized swallowing assessment | day 1 and day 14
  The standardized swallowing assessment was used to assess the improvement of overall swallowing function, it has a maximum score of 46 and a minimum score of 18, with lower scores indicating better swallowing function.

SECONDARY OUTCOMES:
Murray secretion scale | day 1 and day 14
  The severity of Murray secretion scale was measured using a grade of 0-3, patients without obvious saliva accumulation are scored as Murray secretion scale grade 0, whereas patients who had secretions in the laryngeal vestibule at the start of the exam were assigned grade 3.
Rosenbek penetration-aspiration scale | day 1 and day 14
  The highest Rosenbek penetration-aspiration scale score is 8 and the lowest is 1 (1 = no entry of material into the airway; 2 - 5 = penetration of material past the mouse into the supraglottic space and traveling as far as the true vocal folds; 6 - 8 = tracheal aspiration of material below the true vocal folds).
swallowing-quality of life | day 1 and day 14
  Swallowing-quality of life has a score range of 44 - 220, with lower scores indicating poorer swallowing function and poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Xinzhu Rehabilitation Hospital, Xinzhu, Taiwan

IPD SHARING:
Plan to Share IPD: No